CLINICAL TRIAL: NCT05072782
Title: Management of Moderate POstoperative Recurrence in Crohn's Disease: a randoMizEd contROLled Trial of Therapeutic Escalation, the POMEROL Trial. (POMEROL)
Acronym: POMEROL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GT-2021-01
Record Dates: First submitted 2021-08-18; First posted 2021-10-11 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-05

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Rutgeerts score i2; Infliximab CT-P13; Postoperative reccurrence; Ileocolonic resection
MeSH Terms: conditions — Crohn Disease | interventions — CT-P13; 2-mercaptopurine; Methotrexate

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Status quo arm (Other): If the patient received no prophylactic therapy after resection, no treatments will be started.
  If the patient received a prophylactic therapy after resection, the same will be continued at the same dose.
  Interventions: Drug: Immunosuppressors (Thiopurines or Methotrexate)
- Therapy escalation arm (Experimental): Infliximab-CT-P13 will be started with two intravenous infusions of 5 mg per kg bodyweight at week 0 and week 2 and subcutaneous injections of 120 mg every 2 weeks from week 6 onwards.
  Interventions: Drug: Infliximab CT-P13

INTERVENTIONS:
Drug: Infliximab CT-P13 — Stratification 1: Infliximab-CT-P13
  Stratification 2: Infliximab-CT-P13 in combination with immunosuppressors
  Other Names: Remsima
  Arms: Therapy escalation arm
Drug: Immunosuppressors (Thiopurines or Methotrexate) — Stratification 1 : No treatments
  Stratification 2 : Immunosuppressors at same dose
  Arms: Status quo arm

SUMMARY:
Study type : A 30 months, multicentre, open-label strategic randomized controlled trial

Population : Chron's Disease (CD) patients with an i2 endoscopic postoperative recurrence in the year following ileocolonic resection (6-12months after ileocolonic resection).

Treatments :

Stratification at inclusion according to prophylactic therapy.

Patients randomized in 2 arms:

* Status quo arm: if the patient received no prophylactic therapy, no treatment will be started; if the patient received a prophylactic therapy, the same will be continued at the same dose.
* Therapy escalation arm: infliximab-CT-P13 will be started with two intravenous infusions of 5 mg per kg bodyweight at week 0 and week 2 and subcutaneous injections of 120 mg every 2 weeks from week 6 onwards.

Main objective : To evaluate the proportion of CD patients without endoscopic postoperative recurrence (i0-i1) at 12 months in the arm receiving therapy escalation compared to status quo arm in patients having an i2 endoscopic postoperative recurrence 6-12months after ileocolonic anastomosis with restoration of faecal stream.

DETAILED DESCRIPTION:
Number of patients : 360 patients in approximatively 25 sites in France.

Recruitement period : The trial duration for each patients will be 12 months from radomization (18 to 24 months from screening (ie : post-operatively))

Endpoints:

Primary endpoints: Proportion of patients with an i0-i1 modified Rutgeerts score at 12 months.

Secondary endpoints:

* Proportion of patients with an i3-i4 modified Rutgeerts score at 12 months
* Proportion of patients with an i2b-i3-i4 modified Rutgeerts score at 12 months
* Proportion of patients with an i0 modified Rutgeerts score at 12 months
* PRO2 score at 12 months
* Clinical postoperative recurrence within 12 months: average daily SF ≥ 3.5 and average daily AP score ≥ 1.5, AND

  * increased CRP compared to inclusion, at least + 10 mg/l
  * OR increased fecal calprotectin compared to inclusion, at least + 250 μg/g
* Surgical recurrence within 12 months: need for a new ileocolonic resection
* Endoscopic dilatation within 12 months: need for a balloon insufflation at the ileocolonic anastomosis during an ileocolonoscopy when a non-passable stenosis was present in patient having obstructive symptoms (CDOS > 4) before endoscopy
* Time to clinical postoperative recurrence
* Serious adverse events
* Quality of life: EQ5D-5L questionnaire
* Work productivity: Work Productivity and Activity Impairment questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease diagnosed according usual criteria
* Bowel resection with ileocolonic anastomosis performed removing all inflammatory lesions
* Postoperative endoscopy performed between 6 and 12 months after ileocolonic anastomosis reaching the neoterminal ileum (patients who underwent a two stage surgical procedure are also eligible if the endoscopic evaluation is performed 6-12 months after restoration of the fecal stream)
* Moderate endoscopic postoperative recurrence classified i2 according to the Rutgeerts score at 6-12 months, validated by a blinded central reading

Exclusion Criteria:

* Patients with an ostomy
* Ulcerative colitis or IBD type unclassified
* Ileorectal or ileal pouch-anal anastomosis
* Symptoms defined as average daily SF ≥ 3.5 and average daily AP score ≥ 1.5 having started after a free interval without symptoms of at least one month after surgery
* Patients with obstructive symptoms of CD defined by a CDOS > 4
* Patients exposed to infliximab before index surgery with a primary non-response (no clinical effect after 2 infusions at the discretion of the treating gastroenterologist) or history of infusion reactions to infliximab or history of detectable anti-infliximab antibodies
* Patients treated with biological therapy (except for intraocular injections) or an investigational medical product after index surgery
* Patients having started thiopurines or methotrexate more than 6 weeks after ileocolonic anastomosis with restoration of the fecal stream
* Patients in whom not all inflammatory lesions have been removed at index surgery
* Patients with active perianal Crohn's disease
* Patients with a contraindication to infliximab: cancer in the 5 years prior to inclusion excluding non-melanoma skin cancer, active tuberculosis or untreated latent tuberculosis, moderate or severe heart failure, HIV or HBV infection (serology < 6 months), recent live vaccination (within 4 weeks of baseline)
* Pregnant women
* Patients under legal protection or unable to express their consent.
* Patients not affiliated to a health insurance system.
* Patients deprived of liberty by judiciary or administrative decision or hospitalized without consent or admitted in a sanitary or social institution for another reason than research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an i0-i1 modified Rutgeerts score at 12 months. | Month12
  Number of patients with an i0-i1 modified Rutgeerts score at 12 months.

SECONDARY OUTCOMES:
Number of patients with an i3-i4 modified Rutgeerts score at 12 months | Month 12
  Number of patients with an i3-i4 modified Rutgeerts score at 12 months
Proportion of patients with an i2b-i3-i4 modified Rutgeerts score at 12 months | Month 12
  Proportion of patients with an i2b-i3-i4 modified Rutgeerts score at 12 months
Proportion of patients with an i0 modified Rutgeerts score at 12 months | Month 12
  Proportion of patients with an i0 modified Rutgeerts score at 12 months
Patient Reporting Outcome score at 12 months. | Screening, Baseline, week 2, week 6, Month 4, Month 8, Month 12
  Patient Reporting Outcome score at 12 months will be assessed for the evaluation of disease activity (clinical remission).
Clinical postoperative recurrence | Baseline, Month 4, Month 8, Month 12
  Clinical postoperative recurrence within 12 months defined by : Average daily Stool Frequency ≥ 3.5 and average daily Abdominal Pain score ≥ 1.5, AND
  * increased CRP compared to inclusion, at least + 10 mg/l
  * OR increased fecal calprotectin compared to inclusion, at least + 250 μg/g
  Average daily Stool frequency, average daily Abdominal Pain score, CRP and Calprotectin feacal will be combined to report the clinical postoperative recurrence (this outcome is is expressed without units)
Surgical recurrence within 12 months | Baseline, Month 4, Month 8, Month 12
  Surgical recurrence within 12 months defined by need for a new ileocolonic resection. Proportion of surgical recurrence within 12 months
Endoscopic dilatation within 12 months | Baseline, Month 4, Month 8, Month 12
  Endoscopic dilatation within 12 months defined by a need for a balloon insufflation at the ileocolonic anastomosis during an ileocolonoscopy when a non-passable stenosis was present in patient having obstructive symptoms (CDOS > 4) before endoscopy Proportion of endoscopic dilatation within 12 months
Time to clinical postoperative recurrence will be assessed | Baseline, Month 4, Month 8, Month 12
  Time to clinical postoperative recurrence will be assessed
Serious adverse events | Screening, Baseline, Month 4, Month 8, Month 12
  Occurence of Serious Adverse Events
Quality of life: EQ5D-5L questionnaires | Baseline, week 2, week 6, Month 4, Month 8, Month 12
  Quality of life will be assessed with the EQ5D-5L questionnaire
Work productivity and activity impairement questionnaires | Baseline, week 2, week 6, Month 4, Month 8, Month 12
  Work productivity and activity impairement will be assessed with work productivity and activity impairement questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- GETAID, Paris, France